CLINICAL TRIAL: NCT03280589
Title: The Effect of Respiration Rate During Pranayama Practice on the Autonomic Nervous System
Brief Title: Pranayama Practice on the Autonomic Nervous System
Acronym: PYAMA
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: National University of Natural Medicine (Other)
Responsible Party: Principal Investigator, Ryan Bradley, Director, National University of Natural Medicine
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: PYAMA
Record Dates: First submitted 2017-08-09; First posted 2017-09-12 (Actual); Last update posted 2023-03-24 (Actual); Status verified 2023-03

CONDITIONS: Pranayama Effect on Autonomic Nervous System; Respiration Variability Effect on Nervous System
Keywords: Heart Rate Variability; EEG; Respiration
MeSH Terms: conditions — Respiratory Aspiration

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- Sitting Quietly (Active Comparator): Participants will be instructed to sit comfortably in a chair with both feet flat on the floor, hands on their lap or thighs, rest their eyes (closed or slightly open gazed cast down), release tension in the body, remain still, and allow the chair to support them. Instructions will be displayed to them with on-screen video segments while the study personnel helps explains the steps, answers questions, and monitors adherence. There will be 4 five-minute sessions with a one-minute break in between to allow the participant to rest, adjust posture, and answer any questions. The total duration of this session will be approximately 40 minutes.
  Interventions: Other: Sitting Quietly
- Deep Breathing Self Paced (Experimental): Participants will be instructed to sit comfortably in a chair with both feet flat on the floor, hands on their lap or thighs, rest their eyes (closed or slightly open gazed cast down), release tension in the body, remain still, and allow the chair to support them. There will be 4 five-minute sessions with a one-minute break in between to allow the participant to rest, adjust posture, and answer any questions. Instruction will be displayed to them with on-screen video segments while the study personnel helps explains the steps, answers questions, and monitors adherence. The total duration of this session will be approximately 40 minutes.
  Interventions: Other: Deep breathing
- Deep Breathing Externally paced (Experimental): Participants will have an instructional video with auditory queues prompting them to inhale and exhale at 6 bpm (approximately 4 seconds between inhale and exhale). Participants will be instructed to sit comfortably in a chair with both feet flat on the floor, hands on their lap or thighs, rest their eyes (closed or slightly open gazed cast down), release tension in the body, remain still and allow the chair to support them. There will be 4 five-minute sessions with a one-minute break in between to allow the participant to rest, adjust posture, and answer any questions. Instruction will be displayed to them with on-screen video segments while the study personnel helps explains the steps, answers questions, and monitors adherence. The total duration of this session will be approximately 40 minutes.
  Interventions: Other: Deep breathing
- Sheetali/Sheetkali, self-paced: (Experimental): Participant will follow on-screen instructions for Sheetali/Sheetkari with shaped lips/mouth as indicated (i.e., inhaling through the mouth held specific to each practice and exhaling through nostrils), fully filling and emptying the lungs with each breath. In Sheetali, the tongue is allowed to protrude from the mouth at a comfortable distance and rolled into a tube. Following 10 minutes of Sheetali practice, participants will have a one minute rest followed by Sheetkari. In Sheetkari, the tongue is not rolled into a tube; instead, it is rolled up to touch the upper palate. The teeth are then exposed and the lips are kept apart for inhalation and the mouth is closed, tongue is relaxed, and exhalation occurs through the nose. Study personnel will monitor their posture and breathing rate and pause the recording if additional coaching is necessary. The total duration of this session will be approximately 40 minutes.
  Interventions: Other: Sheetali/Sheekari Pranayama; Other: Deep breathing
- Sheetali/Sheetkari, externally-paced (Experimental): The participant will follow on screen instruction for Sheetali/Sheetkari with shaped lips/mouth as indicated, fully filling and emptying the lungs with each breath. The tongue is allowed to protrude from the mouth at a comfortable distance and rolled into a tube. Following 10 minutes of Sheetali practice, participants will have a one-minute rest before continuing. In Sheetkari the teeth are exposed and the lips are kept apart for inhalation and the mouth is closed, tongue is relaxed, and exhalation occurs through the nose. Instruction will be displayed to them with on-screen video segments while the study personnel helps explains the steps, answers questions, and monitors adherence. There will be an auditory queue to prompt the participant to breathe in and out. Study personnel will monitor their posture and breathing rate and pause the recording if additional coaching is necessary.The total duration of this session will be approximately 40 minutes.
  Interventions: Other: Sheetali/Sheekari Pranayama; Other: Deep breathing

INTERVENTIONS:
Other: Sheetali/Sheekari Pranayama — Most pranayama involves (1) sitting quietly, (2) deep breathing (completely filling and emptying the lungs, at a slow/comfortable pace, with awareness), and (3) a specific mouth, tongue, lip and/or body shape, theorized to enhance the effects of the practice. Practitioners of pranayama modulate the cycles of inspiration and expiration, in a way that is theorized to achieve influence over autonomic functions such as heart rate, heart rate variability (HRV), and baroreflex [6]. For example, the manipulation of the tongue and face during Sheetali and Sheetkari pranayama is intended to stimulate parasympathetic nervous system activity and inhibit the sympathetic nervous system.
  Other Names: Pranayama deep breathing
  Arms: Sheetali/Sheetkali, self-paced:; Sheetali/Sheetkari, externally-paced
Other: Sitting Quietly — Participant breaths in their natural way with out instruction
  Arms: Sitting Quietly
Other: Deep breathing — Participant is required to pay attention to each breath
  Arms: Deep Breathing Externally paced; Deep Breathing Self Paced; Sheetali/Sheetkali, self-paced:; Sheetali/Sheetkari, externally-paced

SUMMARY:
The proposed study design will be a randomized, cross-over trial testing different pranayama breathing interventions. Participants (N=40) will perform each of the following five interventions in a randomly assigned order: (1) internal-paced pranayama intervention (Sheetali/Sheetkari for 10 minutes each) (2) internal-paced deep breathing control (3) external-paced pranayama intervention at a rate of 6 bpm (4) external-paced deep breathing at a rate of 6 bpm (5) sitting quietly with no external instruction.

DETAILED DESCRIPTION:
Healthy adult participants (N=40) will be recruited from the general population. Potential participants will contact a study phone line or email expressing their interest, and they will then be contacted in order to schedule a screening telephone interview for an initial assessment of their eligibility. Recruitment will be conducted in the general community using flyers, newspaper advertisements, radio advertisements, and web advertising. NUNM students, faculty, staff and patients will not be specifically targeted for recruitment, although they may see a posted flyer and decide to contact study staff.Screening for potential participants will occur over the phone, using a standardized telephone script and during the first study visit. Prior to all clinical research visits, participants will be called and reminded how to prepare, i.e., avoid extreme physical exercise for one day and refrain from alcohol, caffeinated beverages, and recreational drugs for twelve hours before coming to clinic. The participant will be queried about alcohol, caffeinated beverages, over-the-counter medications, and recreational drugs at the beginning of each visit. If they are not compliant with these instructions, they will be asked to either reschedule their visit until they report compliance or withdraw from the study if compliance is not feasible.

* Height and weight will be measured and recorded and BMI will be calculated (Visit 1 only, if out of range then participant does not meet inclusion criteria and will not be enrolled).
* Heart rate (HR) and blood pressure (BP) will be recorded after the volunteer has been sitting calmly for 5 minutes. The mean of 3 successive recordings with at least 2 minutes between readings will be calculated and recorded as the BP and HR for the visit. (Visit 1 only if out of range then participant does not meet inclusion criteria and will not be enrolled)
* Participants will fill out the pretreatment Mind Body Awareness (visit one and five only) and the Positive Affect Negative Affect Scale (PANAS) questionnaires in order to assess baseline mood.
* Participants will be connected to the ProComp8 infinity Encoder (Thought Technologies) for physiological measurements of EKG (for HR and HRV). For EKG measurement electrodes will be placed on the wrist using adjustable bands. For respiratory measurements thoracic and abdominal sensors will go around the body.
* The order of the following conditions will be randomly assigned (1) self-paced pranayama intervention (Sheetali/Sheetkari consecutively for 10 minutes each) (2) self-paced deep breathing control (3) external-paced pranayama intervention at a rate of 6 bpm (4) external-paced deep breathing at a rate of 6 bpm (5) sitting quietly with no external instruction.
* Before and after measurements will be recorded with the participant's eye open and focused on a on screen image and with eyes closed. This is a common practice in the measurement of EEG due to shifts in Alpha state brain waves when the eyes are closed.
* Each session will follow the pattern below:

  1. Pre- PANAS questionnaire
  2. Intro screen (one activity)

     a. Reviews activities with the participant
  3. Sensor placement

     1. Respiration instructions
     2. EKG instructions
     3. EEG instructions
  4. Eyes open before

     1. Instructions
     2. Measurement
  5. Eyes closed before

     1. Instructions
     2. Measurement
  6. Breathing exercise (Activities unique to each condition with video instructions)

     1. Instructions
     2. Video instructed breath measurement
  7. Eyes open after

     1. Instructions
     2. Measurement
  8. Eyes closed after

     1. Instructions
     2. Measurement
  9. Removal of sensors

     a. Instruction
  10. Post PANAS questionnaire
* Throughout the session participants will be comfortably seated in a chair and instructed to keep their spine erect. The total duration of each HRV measurement will be about 40 minutes: 10 minutes before the practice, 20-minute video with instructions for each condition (broken up into 5 min sections to allow rest), and 10 minutes after the practice.

ELIGIBILITY:
Inclusion Criteria:

* Able to roll tongue into tube (queried over the phone and reassessed at visit 1)
* Age ≥ 25 and ≤ 55 (HRV and other ANS parameters change significantly during the aging process)
* BMI ≥ 18.5 and ≤ 34.9 (Body weight effects HRV and ANS parameters)
* Willing and able to give informed consent
* Able to follow protocol and attend visits
* Able to read and write English
* Able to abstain from over-the-counter painkillers like NSAIDs and allergy medications for 24 hours (Zyrtec and Claritin)

Exclusion Criteria:

* A regular practice of yoga, meditation, and/or breathing more than once a week (Individuals that have conditioned their ANS through yoga, meditation, and breathing exercise may not respond to the breathing condition like the representative population)
* Formal (Yoga Alliance Sanctioned 200h or 500h course or other comparable ) training in yoga, Mindfulness-Based Stress Reduction, transcendental meditation, Qigong, Tai Chi, and/or other forms of meditation/consciousness expansion practices (Individuals that have conditioned their ANS through yoga, meditation, and breathing exercise may not respond to the breathing condition like the representative population)
* A recent cardiovascular event (e.g. myocardial infarction, stroke ≤ six months prior to screening visit), current coronary artery disease, angina, stage III or IV congestive heart failure, or stated history of coronary bypass surgery or heart stent placement
* Presence of a cardiac pacemaker
* History of cardiovascular disease, including heart arrhythmias and prehypertension (systolic BP > 140 mmHg or diastolic BP >90) or hypotension (systolic BP < 90 mmHg or diastolic BP <60)
* Taking prescription drugs that may interfere with heart, nervous, and respiratory rhythms, beta blockers, pain medications, SSRIs, anti-cholinergics, or anxiety medication
* Started or changed the dosage of supplements or medications within the last month
* Open skin rashes and sores that may interfere with placement of sensors
* History of emphysema, chronic bronchitis or bronchiectasis and/or asthma (with FEV1/FVC < 80%) within in the last six months or taking medication to control asthma symptoms
* History of Diabetes type 1 or 2 (> 5 year duration of type 2 diabetes or > 10 years duration of type 1 diabetes (due to the potential for autonomic neuropathy)
* History of or current epilepsy or other seizure disorder(s)
* Current diagnosis of mental illness for which the participant is currently taking prescription medications
* Smoking of tobacco products in a the last 6 months
* Pregnant, nursing, or planning a pregnancy within the next 6 weeks (due to pregnancy-induced changes in HRV
* Presence of any unstable and/or significant medical disorder that would compromise the participant's safety to take part in the trial. Such disorders include any known event that will require beginning new medications and/or prevent adherence to the schedule of study activities over the following 6 weeks
* Chronic hyperventilation (Access by NQ during telephone screen)

Ages: 25 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2017-08-15 (Actual); Primary Completion 2019-05-15 (Actual); Study Completion 2021-07-21 (Actual)

PRIMARY OUTCOMES:
Change in Heart Rate Variability (HRV) | Before and after 20 minutes of breathing excersise
  Analysis of EKG spectra before and after the session

SECONDARY OUTCOMES:
Change in EEG | Before and after 20 minutes of breathing excersise
  Analysis of EEG spectra before and after the session

OTHER OUTCOMES:
Change in PANAS Questionnaire | Before and after 20 minutes of breathing excersise
  Mood Evaluation
Change Mindfullness Questionnaire | Before and after 20 minutes of breathing excersise
  Evaluation of body awareness

CONTACTS AND LOCATIONS:
Locations (1):
- National University of Natural Medicine, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sharpe E, Lacombe A, Sadowski A, Phipps J, Heer R, Rajurkar S, Hanes D, Jindal RD, Bradley R. Investigating components of pranayama for effects on heart rate variability. J Psychosom Res. 2021 Sep;148:110569. doi: 10.1016/j.jpsychores.2021.110569. Epub 2021 Jul 8. PMID 34271528